CLINICAL TRIAL: NCT00003779
Title: A Prospective Randomized Trial for the Comparison of Two BCG Strains (Bacille Calmette-Guerin) in the Prophylaxis of Papollary Bladder Tumors Stage Ta and T1 and Treatment of Carcinoma in Situ
Brief Title: Biological Therapy in Treating Patients With Bladder Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 06/98; SWS-SAKK-06/98 (Other: SAKK); EU-98075 (Other: SAKK)
Record Dates: First submitted 1999-11-01; First posted 2004-03-15 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Bladder Cancer
Keywords: stage 0 bladder cancer; stage I bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BCG-Connaught (Active Comparator)
  Interventions: Biological: Connaught
- BCG Onko-Tice (Active Comparator)
  Interventions: Biological: Tice

INTERVENTIONS:
Biological: Connaught — Compare two strains of BCG
  Arms: BCG-Connaught
Biological: Tice — Compare two strains of BCG
  Arms: BCG Onko-Tice

SUMMARY:
RATIONALE: Biological therapies such as BCG use different ways to stimulate the immune system and stop cancer cells from growing. It is not yet known which type of BCG is more effective for bladder cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of two different types of BCG in treating patients who have bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare two strains of BCG (Connaught vs Tice) in terms of efficacy (yearly relapse rate) and tolerability in patients with Ta or T1 papillary carcinoma of the urinary bladder or carcinoma in situ of the urinary bladder. II. Assess the role of prior exposition to mycobacteria (vaccination/Tbc) for BCG treatment efficacy in these patients. III. Define the role of fever occurrence as a potential indicator for BCG reactivity in these patients. IV. Evaluate the p53 status of the resected tumors and IL-8 secretion into the urine as predictive factors of BCG reactivity in these patients. V. Evaluate disease free interval and disease free survival, time to progression, and overall survival in these patients. VI. Evaluate quality of life in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center, T stage (Ta vs T1 vs CIS), and BCG immunization status (positive, i.e., greater than 10 mm diameter vs negative-indeterminate, i.e., less than 10 mm diameter). All patients undergo complete transurethral resection (TURB) to remove bladder tumors. A Mantoux test is performed. Patients with stage T1 disease undergo a second resection within 2-4 weeks after initial TURB. Patients are randomized to receive either BCG Onko-Tice (arm I) or BCG Connaught (arm II). Both arms receive BCG by catheter beginning 2-14 days after the last TURB. Patients must hold the BCG in the bladder for 2 hours. BCG is instilled once a week for 6 weeks. Quality of life is assessed before randomization, daily during first and last weeks of treatment, every 6 months for the first 2 years, and then annually thereafter. Patients are followed every 6 months for the first 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A minimum of 300 patients will be accrued for this study within 6 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed completely resected T1 or Ta papillary tumors of the urinary bladder TaG2 greater than 2 relapses in 2 years TaG3 unifocal or multifocal Unifocal primary T1G2-3 after a histological tumor-free second resection If multiple/multifocal, worst stage and grade AND/OR Histologically and cytologically confirmed primary or secondary carcinoma in situ of the urinary bladder No persistent T1 disease in second resection No contracted bladder (bladder capacity less than 80 mL) or bladder irritation within past 5 years No urothelial carcinoma of the upper urinary tract or the urethra

PATIENT CHARACTERISTICS: Age: 18 to 90 Performance status: WHO 0-1 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Liver function no greater than 1.5 times upper limit of normal (ULN) Renal: Renal function no greater than 1.5 times ULN Other: Not pregnant or nursing Fertile patients must use effective contraception No other concurrent malignancies except basocellular carcinoma No congenital or acquired immunosuppression (e.g., HIV, leukemia, lymphoma, transplant recipient) No uncontrollable or untreated urinary tract infection No chronic recurring bacterial cystitis

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior BCG therapy Chemotherapy: At least 3 months since prior chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 5 years since prior radiotherapy to the bladder Surgery: See Disease Characteristics Other: No prior tuberculostatic therapy No concurrent local antiseptics or antibiotics

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1998-11; Primary Completion 2001-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Assess role of prior exposition to mycobacteria | 6 weeks

SECONDARY OUTCOMES:
Define role of fever occurrence as potential indicator for BCG reactivity | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: George N. Thalmann, MD, Study Chair — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Inselspital, Bern, Bern, Switzerland

REFERENCES:
- [Result] Rentsch CA, Birkhauser FD, Biot C, Gsponer JR, Bisiaux A, Wetterauer C, Lagranderie M, Marchal G, Orgeur M, Bouchier C, Bachmann A, Ingersoll MA, Brosch R, Albert ML, Thalmann GN. Bacillus Calmette-Guerin strain differences have an impact on clinical outcome in bladder cancer immunotherapy. Eur Urol. 2014 Oct;66(4):677-88. doi: 10.1016/j.eururo.2014.02.061. Epub 2014 Mar 12. PMID 24674149